CLINICAL TRIAL: NCT00179140
Title: The Effects of Protein Supplementation and Resistance Exercise in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Alp Ikizler, Professor, Vanderbilt University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 20064; R01DK045604 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dietary Supplements; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (No Intervention): control period
- 2 (Active Comparator): protein supplementation plus resistance exercise
  Interventions: Drug: nutritional supplementation
- 3 (Active Comparator): protein supplementation only
  Interventions: Drug: nutritional supplementation; Behavioral: exercise

INTERVENTIONS:
Drug: nutritional supplementation — oral administration of protein supplement (Nepro) during hemodialysis; every other day, 3 days per week for 6 months; Nepro is a lactose-free formula that contains a total of 960 kilocalories: 132.8 kilocalories from protein, 412.8 kilocalories from carbohydrates, and 412.8 kilocalories from fat
  Arms: 2; 3
Behavioral: exercise — either before or during hemodialysis, patients will perform a leg press exercise; every other day, 3 days per week, for 6 months
  Arms: 3

SUMMARY:
The objective of this study is to determine how protein supplementation, with or without exercise, affects functional capacity, strength, body composition, and physical activity in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* On hemodialysis for more than 3 months, on a thrice weekly hemodialysis program;
* Adequately dialyzed (Kt/V > 1.4).
* Age > 18 years old.
* Properly functioning AV Graft

Exclusion Criteria:

* Patients unable to perform exercise due to cardiovascular disease, osteoarthritis, etc.
* Pregnant women.
* Severe unstable underlying disease besides commonly associated with ESRD. Cardiac patients that are stable will be included.
* Patients hospitalized within the last month prior to the study.
* Patients will not perform the MRI if contraindication as determined using the VUMC MRI Procedure Screening Form (attached) or prior claustrophobic reaction in an MRI scanner.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2002-11; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
increase in lean body mass | 13 months

SECONDARY OUTCOMES:
improve physical functioning | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Alp Ikizler, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Bernier-Jean A, Beruni NA, Bondonno NP, Williams G, Teixeira-Pinto A, Craig JC, Wong G. Exercise training for adults undergoing maintenance dialysis. Cochrane Database Syst Rev. 2022 Jan 12;1(1):CD014653. doi: 10.1002/14651858.CD014653. PMID 35018639
- [Derived] Mah JY, Choy SW, Roberts MA, Desai AM, Corken M, Gwini SM, McMahon LP. Oral protein-based supplements versus placebo or no treatment for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2020 May 11;5(5):CD012616. doi: 10.1002/14651858.CD012616.pub2. PMID 32390133